CLINICAL TRIAL: NCT00325208
Title: Feeding Bottle Design, Milk Intake and Infant Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06NT01
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Healthy Infants

INTERVENTIONS:
Device: partial-vacuum milk bottle
Device: anti-vacuum milk bottle

SUMMARY:
It is increasingly recognised that rapid growth in infancy may be associated with a greater risk of cardiovascular disease later in life. This trial will investigate whether the use of infant feeding bottles with different designs influences the milk intake and growth of infants. We will compare the growth of bottle-fed infants with that of a breast-fed reference group.

ELIGIBILITY:
Inclusion Criteria:

* healthy term infants birth weight >2.50kg, gestational age >37 weeks

Exclusion Criteria:

-

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152
Dates: Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fewtrell, Principal Investigator — Institute of Child Health
Locations (3):
- United Kingdom (3):
  - Hillingdon hospital, London
  - Northwick Park Hospital, London
  - The Institute of Child health, London

REFERENCES:
- [Derived] Fewtrell MS, Kennedy K, Nicholl R, Khakoo A, Lucas A. Infant feeding bottle design, growth and behaviour: results from a randomised trial. BMC Res Notes. 2012 Mar 16;5:150. doi: 10.1186/1756-0500-5-150. PMID 22424116